CLINICAL TRIAL: NCT03806764
Title: Assessing the Impact and Complications of Cytomegalovirus (CMV) Reactivation in a Multi-site Study of Allogeneic Haematopoietic Stem Cell Transplant Recipient
Brief Title: Cytomegalovirus (CMV) Reactivation in Allogeneic HSCT Recipient
Acronym: CReSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Melbourne Health (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other); Western Sydney Local Health District (Other); Walter and Eliza Hall Institute of Medical Research (Other); Austin Hospital, Melbourne Australia (Other)
Responsible Party: Principal Investigator, Monica Slavin, Infectious Diseases Physician, Melbourne Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CReSCT
Record Dates: First submitted 2019-01-07; First posted 2019-01-16 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cytomegalovirus Infections; Haematological Malignancy; Organ or Tissue Transplant; Complications; Immune Suppression
Keywords: Cytomegalovirus; CMV; Reactivation; HSCT; Stem cell transplant; allogeneic; immunosuppression; viral infection
MeSH Terms: conditions — Cytomegalovirus Infections; Hematologic Neoplasms; Virus Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The study consists of a retrospective and a prospective parts on patients developing CMV infection post allogeneic haematopoeitic stem cell transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Retrospective study (No Intervention): Medical records of 250 allo-HSCT recipients will be evaluated retrospectively to determine the incidence and clinical outcomes of CMV viremia post HSCT, including both the direct (CMV disease) and indirect (such as invasive fungal infection, other viral infections, bacterial infection) effects on clinical outcomes.
- Prospective study (Other): 120 recipients of allo-HSCT will be recruited into the prospective part of the study. Participants will be reviewed pre-transplant, 6, 12, 24 and 52 weeks following HSCT during routine clinical visits. clinical assessment will be made such as CMV viremia, transplant related complications and current medications.
  Participants who are at high risk of CMV will have study blood sampling taken to assess immune functions
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood sampling from prospective study participants will be taken for immune functions measurements
  Arms: Prospective study

SUMMARY:
This study consists of two parts: 1) Part 1, a retrospective part on 250 consecutive patients following allogeneic haematopoietic stem cell transplant (allo-HSCT) at the Royal Melbourne Hospital from 2012 to 2017, inclusive, and 2) Part 2, a prospective part on 120 allo-HSCT patients from 4 sites in Australia: the Royal Melbourne Hospital, Peter MacCallum Cancer Centre, Austin Hospital, and Westmead Hospital.

In Part 1, medical records of allo-HSCT recipients will be evaluated to determine the incidence and clinical outcomes of CMV viremia post HSCT, including both the direct (CMV disease) and indirect (such as invasive fungal infection, other viral infections, bacterial infection) effects on clinical outcomes.

In Part 2, allo-HSCT participants at risk of CMV disease will be assessed to determine the association of host CMV-specific immunity with clinical management and outcomes over one year post allo-HSCT.

The overall aims of the study are to establish if CMV infection in allo-HSCT patients are associated with poor clinical outcomes; and whether measurement of immunological functions could provide an early indicator to identify patients at risk and appropriate timing for initiation of CMV treatment.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) infection is recognised as one of the most common and important infectious complication of allogeneic haematopoietic stem cell transplantation (allo-HSCT). Despite the serious clinical implications of CMV reactivation, there is a paucity of data informing clinicians on how to best identify 'at risk' patients, timely commencement of management of the infection.

This study consists of two parts: 1) Part 1, a retrospective part, and 2) Part 2, a prospective part.

In Part 1, a retrospective cohort of 250 recipients of allo-HSCT at the Royal Melbourne Hospital will be reviewed. The study period will be between January 2012- December 2017, inclusive. The follow up period will be 6 months from the day of transplantation (ie. day 0 to 180). Data on patient demographics (age, sex, ethnicity), primary indication for transplantation, donor type (match, unmatched, minor mismatch, related or unrelated), graft source (stem cell, bone marrow, umbilical cord) conditioning regimen (myeloablative reduced intensity conditioning), graft versus host disease (GVHD) prophylaxis eg. T-cell depletion, days to neutrophil recovery, occurrence of acute and chronic GVHD and the therapy for GVHD (including steroid intensity, use of ATG etc.), associated bacterial and fungal infections, relapse and mortality, will be collected for analyses. CMV-negative patients will be used as control for economic comparisons.

In Part 2, 120 recipients of allo-HSCT will be recruited from 4 Australian hospitals (the Royal Melbourne Hospital, Austin Hospital, Peter MacCallum Cancer Centre, and Westmead Hospital). Participants will be reviewed pre-transplant, 6, 12, 24 and 52 weeks following HSCT during routine clinical visits. Clinical assessment will be made such as CMV viremia, transplant related complications and current medications. In addition, participants who are at high risk of CMV will have study bloods taken to assess immune functions with Quantiferon-CMV®, Quantiferon-Monitor® assay, CMV Elispot, peripheral blood mononuclear cells (PBMCs) and plasma for storage at time-points of 0, 6 and 12 weeks +/- 2 weeks after commencing anti-CMV treatment. The Quantiferon-Monitor® assay will be performed at the additional time points of 4, 18 and 26 weeks following HSCT.

ELIGIBILITY:
Inclusion Criteria:

* For the retrospective cohort, all 250 consecutive allo-HSCT patients between 2012 to 2017 at the Royal Melbourne Hospital will be included, with CMV-negative patients acting as controls for economic comparisons.
* For the prospective cohort, patients undergoing allo-HSCT, at risk of CMV disease (D+/R+, D-/R+ D+/R-), and able to provide informed consent.

Exclusion Criteria:

* For the retrospective cohort, no exclusion is set.
* For the prospective cohort, patients who has CMV disease at the time of enrolment and patients who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and outcome of CMV viremia | 250 retrospective cases of HSCTduring 2012 to 2017, inclusive, will be reviewed from the day of transplant to 6 months post transplant.
  The incidence and outcome of clinically relevant CMV viremia post HSCT will be assessed
Host CMV-specific T cell immunity and related clinical outcomes | 52 weeks following HSCT
  Host CMV-specific T cell immunity status of 120 participants will be assessed prospectively against CMV related clinical outcomes to establish if correlations exist

SECONDARY OUTCOMES:
Low level CMV viremia | 250 retrospective cases of HSCTduring 2012 to 2017, inclusive, will be reviewed from the day of transplant to 6 months post transplant.
  Association of low level CMV viremia and the subsequent clinical outcomes
Economic cost for managing CMV infection | 250 retrospective cases of HSCTduring 2012 to 2017, inclusive, will be reviewed from the day of transplant to 6 months post transplant.
  The economic cost attributable to managing CMV infection and CMV disease will be evaluated to provide a picture of health economics of the infection
CMV viral load for initiation of treatment | 52 weeks following HSCT
  CMV viral load will be assessed to determine an appropriate trigger to initiate treatment for CMV viremia
Correlation of host T cell function and risk of CMV infection | 52 weeks following HSCT
  Association of low or inadequate global immune function (T-cell and TLR7 responses) will be correlated with an increased risk of developing CMV infection post HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Monica Slavin, MBBS FRACP, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Parkville, Victoria, Australia